CLINICAL TRIAL: NCT04535583
Title: Harnessing Digital Health to Understand Clinical Trajectories of Opioid Use Disorder
Acronym: D-TECT
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Drug Abuse Treatment Clinical Trials Network (Network); Dartmouth College (Other); Kaiser Permanente (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa A. Marsch, Professor, Dartmouth-Hitchcock Medical Center
Other Study IDs: CTN-0084-A2; UG1DA040309 (NIH); UG1DA040314 (NIH)
Record Dates: First submitted 2020-08-03; First posted 2020-09-02 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Opioid-use Disorder
Keywords: Opioid Use Disorder; Digital Health; Substance Use Disorder; Social Media
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EMA plus passive sensing: Participants will be responding to up to 3 ecological momentary assessments per day plus carrying a smartphone and wearing a smartwatch. Both the smartphone and smartwatch will passively collect sensor data continuously.

SUMMARY:
The main objective of the study is to evaluate the feasibility of utilizing digital health technology with opioid use disorder (OUD) patients as measured by a 12-week period of continuous assessment using smartphone surveys and digital sensing. In addition, we will examine the utility of 3 types of digital data (Ecological Momentary Assessment (EMA); Digital sensing; and social media data) in predicting OUD treatment retention and buprenorphine medication adherence.

DETAILED DESCRIPTION:
This is an observational study designed to (1) evaluate the feasibility and utility of digital health technology in a Medication for Opioid Use Disorder (MOUD) treatment population, and (2) capitalize on the availability of Electronic Health Record (EHR) data to relate passive and active sensing data to treatment retention and medication adherence.

Eligible participants are identified through EHR records, sent an invitational letter through secure message, and then called to recruit and screen. Following verbal consent to screen, research staff will perform a screening assessment over the phone/video to determine preliminary study eligibility prior to scheduling the baseline phone/video appointments. Following electronic signed informed consent, participants will be asked to complete an interviewer administered Baseline assessment. In addition to the screening and baseline assessments, the participants will be asked to wear a smartwatch and carry a smartphone continuously for a period of 12 weeks. Smartphone and smartwatch data will be passively collected. In addition, participants will be prompted to respond to questions through a smartphone (i.e., Ecological Momentary Assessment (EMA)) 3 times daily for 12 weeks. In addition to the EMA prompts, individuals will be asked to self-initiate EMAs if substance use occurred.

After the 12-week active study phase, participants will be asked to complete a follow-up phone/video appointment.

EHR and medical claims data will be extracted 16 weeks after study completion (data will be collected 12 months prior to EMA start through 12 weeks after EMA start).

For those who consent to the optional social media component, social media data will be downloaded by the participant directly from the social media platform to a secure server using a remote desktop at the beginning of the study and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have been active in Kaiser outpatient buprenorphine treatment for OUD for the past 2 weeks (determined at screening);
2. Be ≥18 years old (determined at screening);
3. Be able to understand English (determined at screening);
4. Be available to participate in the full duration of the study (12 weeks) (determined at screening);
5. Have an active email account and willing to provide the email address to researchers (determined at screening);
6. Permit researchers to access personal electronic health record (EHR) and medical claims data (determined at screening);
7. Be willing to carry and use personal or study provided smartphone for 12 weeks (determined at screening); and
8. Be willing to wear a smartwatch continuously (except during pre-defined activities such as showering) for 12 weeks (determined at screening).

Exclusion Criteria:

1. Are unwilling or unable to provide informed consent (determined during the Consent process and during Consent Quiz); and
2. Are currently in jail, prison or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities (determined by Prisoner Status Assessment at each study visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is recruiting individual who are active in medication treatment for opioid use disorder (MOUD) with buprenorphine for at least 2 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Marsch, PhD, Principal Investigator — Dartmouth College; Cynthia Campbell, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available by the Principal Investigators upon request.
Supporting Information: Study Protocol
Time Frame: Data will be available after the completion of the study and data lock.
Access Criteria: Prior to receiving any study data, researchers/institutions will need to enter into a data sharing agreement with the institution(s) providing the de-identified study data.

REFERENCES:
- [Derived] Marsch LA, Chen CH, Adams SR, Asyyed A, Does MB, Hassanpour S, Hichborn E, Jackson-Morris M, Jacobson NC, Jones HK, Kotz D, Lambert-Harris CA, Li Z, McLeman B, Mishra V, Stanger C, Subramaniam G, Wu W, Campbell CI. The Feasibility and Utility of Harnessing Digital Health to Understand Clinical Trajectories in Medication Treatment for Opioid Use Disorder: D-TECT Study Design and Methodological Considerations. Front Psychiatry. 2022 Apr 29;13:871916. doi: 10.3389/fpsyt.2022.871916. eCollection 2022. PMID 35573377

RESULTS

PARTICIPANT FLOW:
Groups:
- EMA Plus Passive Sensing (Social Media Optional): Participants will be responding to up to 3 ecological momentary assessments per day plus carrying a smartphone and wearing a smartwatch. Both the smartphone and smartwatch will passively collect sensor data continuously. Participation in the social media data collection portion of the study was optional. Participants with social media accounts could consent to share their social media data with the study team.
Period: Overall Study
Arm/Group | EMA Plus Passive Sensing (Social Media Optional)
Started | 65
Completed | 62
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | EMA Plus Passive Sensing (Social Media Optional)
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (13.3)
Sex/Gender, Customized [Number; unit: participants]
  Male | 32
  Female | 31
  Other | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 46
  Non-white/more than one race | 19
  Hispanic/Latino/of Spanish origin | 14
  Non-Hispanic | 51
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Smartphone Sensor Data
Description: The percentage of days carried the smartphone at least 8 hours per day.
Time Frame: 84 days (or 12-weeks)
Population: 62 out of the 65 participants completed the baseline visit and received the study smartphone or had the study app setup on their personal smartphone to contribute passive data via smartphone.
Measure: Mean (95% Confidence Interval); unit: mean percentage of days
Arm/Group | EMA Plus Passive Sensing (Social Media Optional)
Number analyzed (Participants) | 62
mean percentage of days | 94.2 [90.8 to 97.6]

2. Secondary Outcome: Social Media Data
Description: The percentage of participants who consented to download social media data.
Time Frame: At baseline
Population: 49 out of 56 participants had social media accounts. Therefore, the denominator used to determine the percentage of participants who consented to download social media data was the total number of participants with social media accounts.
Measure: Count of Participants; unit: Participants
Arm/Group | EMA Plus Passive Sensing (Social Media Optional)
Number analyzed (Participants) | 56
Participants | 49

3. Secondary Outcome: The Number of Ecological Momentary Assessments (EMA) With Response
Description: The response rate to Ecological Momentary Assessment prompts during the 12-week study phase. The EMA Response Rate for each participant is the number of EMAs responded to over the last 83 days of the study (up to 249 responses [83 days X 3 EMA]) (yields a percentage). The total mean EMA response rate was based on the EMA response rate (percentage) across all participants in the study (N=62).
Time Frame: up to 3 times per day for 84 days (or 12-weeks)
Population: 62 out of the 65 participants completed the baseline visit and received the study smartphone or had the study app setup on their personal smartphone to respond to ecological momentary assessments.
Measure: Mean (95% Confidence Interval); unit: mean percentage of EMA response rate
Arm/Group | EMA Plus Passive Sensing (Social Media Optional)
Number analyzed (Participants) | 62
mean percentage of EMA response rate | 70.0 [63.5 to 81.4]

4. Secondary Outcome: Smartwatch Sensor Data
Description: The percentage of days wore the smartwatch at least 18 hours per day.
Time Frame: 84 days (or 12-weeks)
Population: 62 out of the 65 participants completed the baseline visit and received the study smartwatch to contribute passive data via smartwatch.
Measure: Mean (95% Confidence Interval); unit: Mean percentage of days
Arm/Group | EMA Plus Passive Sensing (Social Media Optional)
Number analyzed (Participants) | 62
Mean percentage of days | 73.7 [67.7 to 79.7]

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | EMA Plus Passive Sensing (Social Media Optional)
All-Cause Mortality (participants affected / at risk) | 1/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 5/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMA Plus Passive Sensing (Social Media Optional) (N=65)
Suicidal Ideation (Psychiatric disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT04535583/Prot_SAP_000.pdf